CLINICAL TRIAL: NCT05536973
Title: A Multi-Center, Randomized, Double-Masked Phase 2 Study to Assess Safety and Efficacy of ADVM-022 (AAV.7m8-aflibercept) in Anti-VEGF Treatment-Experienced Patients With Neovascular (Wet) Age-related Macular Degeneration (nAMD) [LUNA]
Brief Title: Safety and Efficacy of ADVM-022 in Treatment-Experienced Patients With Neovascular Age-related Macular Degeneration [LUNA]
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADVM-022-11
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: Aflibercept; Best Corrected Visual Acuity; Adverum; ADVM; ADVM-022; ADVM-022-11; Age-related macular degeneration; Wet macular degeneration; Wet AMD; Choroidal neovascularization; CNV; AAV.7m8; Anti-VEGF therapy; Gene therapy; Blindness; AAV; AAV vector; nAMD; wAMD; Eye disease; Eye diseases
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Choroidal Neovascularization; Blindness; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Experimental): A single intravitreal injection of ADVM-022 2E11 vg/eye
  Interventions: Genetic: ADVM-022
- Dose 2 (Experimental): A single intravitreal injection of ADVM-022 6E10 vg/eye
  Interventions: Genetic: ADVM-022

INTERVENTIONS:
Genetic: ADVM-022 — A single IVT injection of 2E11 vg/eye ADVM-022 dose in combination with one (1) of four (4) corticosteroid treatment regimens
  Arms: Dose 1
Genetic: ADVM-022 — A single IVT injection of 6E10 vg/eye ADVM-022 dose in combination with one (1) of four (4) corticosteroid treatment regimens
  Arms: Dose 2

SUMMARY:
Neovascular or wet age-related macular degeneration (nAMD) is a degenerative ocular disease associated with the infiltration of abnormal blood vessels in the retina from the underlying choroid layer and is a leading cause of blindness in patients over 65 years of age. The abnormal angiogenic process in nAMD is stimulated and modulated by vascular endothelial growth factor (VEGF). Treatment of nAMD requires frequent intravitreal (IVT) injections of VEGF inhibitors (anti-VEGF) administered every 4-16 weeks. ADVM-022 (AAV.7m8-aflibercept) is a gene therapy product being developed for the treatment of nAMD and offers the potential for sustained intraocular expression of aflibercept following a single IVT injection. ADVM-022 is designed to reduce the current treatment burden which often results in undertreatment and vision loss in patients with nAMD receiving anti-VEGF therapy in clinical practice.

DETAILED DESCRIPTION:
This Phase 2, multi-center, randomized, double-masked, parallel group study is designed to evaluate the safety, tolerability, and efficacy of a single IVT injection of ADVM-022 at one of two doses (2 × 10^11 vg/eye [2E11] or 6 × 10^10 vg/eye [6E10]) accompanied by one of four prophylactic corticosteroid treatment regimens.

Anti-VEGF treatment-experienced study participants meeting the eligibility criteria that will be randomized between the 2E11 vg/eye and 6E10 vg/eye ADVM-022 doses each with 4 prophylaxis arms for a total of 8 treatment arms, and only one eye per study participant will be selected as the study eye.

Safety, tolerability, and efficacy will be evaluated for a period of approximately 5 years from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, ≥ 50 years of age
* Willing and able to provide written, signed informed consent for this study
* Demonstrated a meaningful response to anti-VEGF therapy
* Participants must be under active anti-VEGF treatment for wet AMD and received a minimum of 2 injections within 4 months prior to screening for the treatment of choroidal neovascularization secondary to nAMD in the study eye
* Vision of the study eye at Baseline: BCVA in the range of 25 - 83 ETDRS letters, inclusive (approximate Snellen equivalent visual acuity range of 20/25 - 20/320)
* Vision of the non-study eye at Baseline: BCVA ≥ 35 ETDRS letters (approximate Snellen equivalent of 20/200 or better)

Exclusion Criteria:

* Any condition that could affect the interpretation of results or render the participant at high risk of treatment complications in the opinion of the Investigator
* Ocular or periocular infection or intraocular inflammation in either eye within 1 month prior to or at the Randomization Visit (Day -7)
* Uncontrolled diabetes or HbA1c ≥ 7.0 %
* History or evidence of significant uncontrolled concomitant disease within 6 months of the Screening visit
* Any history of ongoing bleeding disorders or INR >3.0
* History or evidence of macular or retinal disease other than nAMD
* History or evidence of retinal detachment or retinal pigment epithelium rip/tear
* Uncontrolled ocular hypertension or glaucoma
* Prior treatment with photodynamic therapy or retinal laser for the treatment of nAMD
* Any history of vitrectomy or any other vitreoretinal surgery
* Prior treatment with gene therapy at any time or any non-gene therapy investigational treatment or medical device in the study eye within 3 months of the Screening Visit or 5 half-lives of the investigational medicinal product

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and non-ocular adverse events | Up to Week 52
  Incidence of ocular and non-ocular adverse events
Severity of ocular and non-ocular adverse events | Up to Week 52
  Severity of ocular and non-ocular adverse events
Mean change in best corrected visual acuity (BCVA) from Baseline | Baseline up to Week 52
  BCVA measured by Early Treatment Diabetic Retinopathy Study (ETDRS)

SECONDARY OUTCOMES:
Percentage of participants from Baseline who lose/gain at least 5, 10 or 15 letters in BCVA | Baseline up to 5 years
  BCVA measured by ETDRS
Mean change in BCVA from Baseline | Baseline up to 5 years
  BCVA measured by ETDRS
Percentage of participants who are supplemental aflibercept injection-free | Baseline up to 5 years
  Supplemental anti-VEGF treatments required post therapy
Percent reduction in annualized anti-VEGF injections | Baseline up to 5 years
  Supplemental annualized anti-VEGF treatments required post therapy to the year prior
Mean change in Central Subfield Thickness (CST) from Baseline | Baseline up to 5 years
  To evaluate the effect of ADVM-022 on CST
Percentage of participants without CST fluctuations | Baseline up to 5 years
  To evaluate the effect of ADVM-022 on CST
Mean number of CST fluctuations from Baseline | Baseline up to 5 years
  To evaluate the effect of ADVM-022 on CST
Percentage of participants without post-prophylactic inflammation | Baseline up to 5 years
  To assess the long-term safety and tolerability of a single IVT injection of ADVM-022
Incidence of ocular and non-ocular adverse events | Up to 60 months
  To assess the long-term safety and tolerability of a single IVT injection of ADVM-022
Severity of ocular and non-ocular adverse events | Up to 60 months
  To assess the long-term safety and tolerability of a single IVT injection of ADVM-022

CONTACTS AND LOCATIONS:
Overall Officials: Adam Turpcu, PhD, Study Director — Adverum Biotechnologies, Inc.
Locations (39):
- United States (34):
  - Adverum Clinical Site 178, Phoenix, Arizona
  - Adverum Clinical Site 126, Phoenix, Arizona
  - Adverum Clinical Site 159, Tucson, Arizona
  - Adverum Clinical Site 100, Beverly Hills, California
  - Adverum Clinical Site 172, Encino, California
  - Adverum Clinical Site 169, Fullerton, California
  - Adverum Clinical Site 170, Pasadena, California
  - Adverum Clinical Site 174, Poway, California
  - Adverum Clinical Site 164, Riverside, California
  - Adverum Clinical Site 166, Sacramento, California
  - Adverum Clinical Site 175, Santa Barbara, California
  - Adverum Clinical Site 116, Lakewood, Colorado
  - Adverum Clinical Site 165, Waterford, Connecticut
  - Adverum Clinical Site 124, Deerfield Beach, Florida
  - Adverum Clinical Site 176, Fort Lauderdale, Florida
  - Adverum Clinical Site 168, Jacksonville, Florida
  - Adverum Clinical Site 149, ‘Aiea, Hawaii
  - Adverum Clinical Site 167, Detroit, Michigan
  - Adverum Clinical Site 161, Royal Oak, Michigan
  - Adverum Clinical Site 163, Southaven, Mississippi
  - Adverum Clinical Site 177, Omaha, Nebraska
  - Adverum Clinical Site 119, Reno, Nevada
  - Adverum Clinical Site 146, Cherry Hill, New Jersey
  - Adverum Clinical Site 171, Teaneck, New Jersey
  - Adverum Clinical Site 122, West Columbia, South Carolina
  - Adverum Clinical Site 144, Rapid City, South Dakota
  - Adverum Clinical Site 101, Nashville, Tennessee
  - Adverum Clinical Site 123, Abilene, Texas
  - Adverum Clinical Site 154, Austin, Texas
  - Adverum Clinical Site 108, Bellaire, Texas
  - Adverum Clinical Site 162, McAllen, Texas
  - Adverum Clinical Site 151, San Antonio, Texas
  - Adverum Clinical Site 107, The Woodlands, Texas
  - Adverum Clinical Site 152, Morgantown, West Virginia
- France (3):
  - Adverum Clinical Site 502, Nantes, Loire-Atlantique
  - Adverum Clinical Site 501, Lyon, Rhône
  - Adverum Clinical Site 500, Créteil, Val-de-Marne
- United Kingdom (2):
  - Adverum Clinical Site 600, London
  - Adverum Clinical Site 601, Oxford

IPD SHARING:
Plan to Share IPD: Undecided